CLINICAL TRIAL: NCT03304041
Title: Efficacy of Low-FODMAPs Dietary Therapy Versus Traditional Dietary Advice for Diarrhea-predominant Irritable Bowel Syndrome in China - A Prospective Randomized Controlled Trial
Brief Title: Efficacy of Low-FODMAPs Dietary Therapy for Irritable Bowel Syndrome in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Zhejiang Academy of Agricultural Sciences (Unknown); University of Michigan (Other); Klinik Arlesheim (Other)
Responsible Party: Principal Investigator, DAI Ning, Director of Gastroenterology department, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170116-2
Record Dates: First submitted 2017-07-20; First posted 2017-10-06 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Irritable Bowel Syndrome; Diet Modification
Keywords: low-FODMAP; Irritable Bowel Syndrome; stool fermentation; Breath test
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-FODMAPs diet (Experimental): The low-FODMAPs diet(LFD) aims to keep oligosaccharides, fructose in excess of glucose, and polyol content at less than 0.5 g each per serving based on previously published data.
  low-FODMAPs diet therapy for 3 weeks
  Interventions: Dietary Supplement: low-FODMAPs diet
- Traditional dietary advice (Placebo Comparator): Traditional dietary advice (TDA) will focus more on how and when to eat rather than on what foods to ingest . Patients will be instructed to regularly eat, never too much or too little, never to be hungry or too full; to eat in peace and to chew thoroughly; reduce intake of fatty, spicy food, fiber, coffee and alcohol during the intervention period
  Traditional dietary advice for 3 weeks
  Interventions: Dietary Supplement: Traditional dietary advice

INTERVENTIONS:
Dietary Supplement: low-FODMAPs diet — The low-FODMAPs diet(LFD) aims to keep oligosaccharides, fructose in excess of glucose, and polyol content at less than 0.5 g each per serving based on previously published data.
  low-FODMAPs diet therapy for 3 weeks
  Arms: low-FODMAPs diet
Dietary Supplement: Traditional dietary advice — Traditional dietary advice(TDA) will focus more on how and when to eat rather than on what foods to ingest . Patients will be instructed to regularly eat, never too much or too little, never to be hungry or too full; to eat in peace and to chew thoroughly; reduce intake of fatty, spicy food, fiber, coffee and alcohol during the intervention period
  traditional dietary advice for 3 weeks
  Arms: Traditional dietary advice

SUMMARY:
The primary aim of our study is to carry out a randomized trial to evaluate the efficacy of low-FODMAPs dietary therapy compared to conventional therapy for IBS patients recruited from tertiary hospitals in China. Secondary aims of this research include an analysis of clinical, physiological and microbiological factors that may predict IBS patient response to this dietary intervention.

DETAILED DESCRIPTION:
Visit 1：Enrollment & Screening & Run-in period Patients who meet the inclusion criteria will be asked to complete IBS Baseline Assessment Questionnaires according to Rome III.Subjects that meet the criteria will receive verbal and written information about the study and provide written informed consent. After meeting with the dietitian and physician who will provide instructions, they will be asked to complete Combined Nutrient and Lactulose Breath Test.[16] Additionally, a baseline food and symptom diary will be completed in a (minimum) 14 day run-in period after breath test (the first 48hr after the breath test will not be included in this analysis). This diary record prior to the intervention will document baseline symptom severity and capture the habitual diet of IBS patients.

Visit 2: Randomization & Intervention. After the run-in period, patients will come back to the clinic to receive dietary instruction ahead of starting the intervention. At the same visit subjects will provide fresh stool for fermentation analysis (including short chain fatty acids and pressure detection) and blood for cytokines analysis. Subjects will then be randomly assigned to either low FODMAP diet (LFD) group or traditional dietary advice for IBS (TDA) group by computer-generated random number table. Participants will receive food instructions by a dietitian, according to their assignment. Throughout the study, only the dietitian will be aware of the assignment of the intervention given. Both diet therapy will last for 3 weeks, and all the subjects are instructed to complete daily food and symptom diary through a provided booklet. IBS Symptoms Severity Scores (IBS-SSS) is evaluated every week and the dietitian who is not aware of the allocation will make a telephone follow-up to assess patient adherence.

Visit 3: End of treatment & Follow-up. After 3 weeks of intervention, the participants will attend a follow-up appointment and complete the IBS Post-Intervention Assessment Questionnaires. Fresh stools and blood are recollected at this visit to evaluate for possible change in gut microbiota and cytokines after diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* Meet Rome Rome III criteria for IBS-D.
* All these patients should have no abnormality in blood, stool analysis or colonoscopy within the previous 2 years.
* No GI alarm symptoms.

Exclusion Criteria:

* Presence of a severe cardiac, hepatic, nephritic, neurologic disease.
* Presence of mental disorders caused by schizophrenia, organic brain disorder or physical disease.
* Other comorbid medical conditions (eg.unstable diabetes, unstable thyroid disease).
* Previous abdominal surgery except appendectomy or hysterectomy.
* Pregnant or lactating women.
* Use of probiotics, prebiotics, lactulose, antidiarrheal agents or bowel preparation within the 4 weeks prior to the study.
* Participation in any other form of dietary therapy within the 4 weeks prior to the study.
* Difficulties in communication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Compare response to diet intervention between different groups. | three weeks
  Primary endpoint will be response to 3-week of diet intervention defined by shows >50 point reduction in IBS-SSS between baseline and post-intervention scores. The proportion of responders who met primary endpoint in each group will be compared.

SECONDARY OUTCOMES:
Improvement in abdominal pain between different groups. | Three weeks
  Compare improvement about abdominal pain during 3-week intervention period between different groups according to Food and Drug Administration (FDA) individual composite end point (≥30% reduction in mean daily abdominal pain score).
Improvement in stool consistency between different groups. | Three weeks
  Compare improvement about stool consistency during 3-week intervention period between different groups according to Food and Drug Administration (FDA) individual composite end point (a decrease in mean daily Bristol Stool Score (BSS) value of ≥1 compared with baseline for any 2 weeks of the intervention period).
Compare changes from baseline in abdominal pain score between different groups. | Every week, last for three weeks
  Compare group changes from baseline in abdominal pain score，averaged over each treatment week for total three weeks.
Compare changes from baseline in abdominal frequency between different groups. | Every week, last for three weeks
  Compare group changes from baseline in abdominal frequency, averaged over each treatment week for total three weeks.
Compare changes from baseline in bloating score between different groups. | Every week, last for three weeks
  Compare group changes from baseline in bloating score, averaged over each treatment week for total three weeks.
Compare changes from baseline in excessive wind score between different groups. | Every week, last for three weeks
  Compare group changes from baseline in excessive wind score, averaged over each treatment week for total three weeks.
Compare changes from baseline in stool consistency between different groups. | Every week, last for three weeks
  Compare group changes from baseline in stool consistency as measured by BSS, averaged over each treatment week for total three weeks..
Compare changes from baseline in stool frequency between different groups. | Every week, last for three weeks
  Compare group changes from baseline in stool frequency, averaged over each treatment week for total three weeks.
Compare changes from baseline in urgency score between different groups. | Every week, last for three weeks
  Compare group changes from baseline in urgency score, averaged over each treatment week for total three weeks.
Compare changes from baseline in incomplete defecation score between different groups. | Every week, last for three weeks
  Compare group changes from baseline in incomplete defecation score, averaged over each treatment week for total three weeks.
Compare changes from baseline in quality of life between different groups. | Three weeks
  Compare group changes between baseline and post-intervention(3 weeks later) about quality of life evaluated by IBS-QOL.
Compare changes from baseline in mental health between different groups. | Three weeks
  Compare group changes between baseline and post-intervention(3 weeks later) about mental health evaluated by GAD-7 and PHQ-9.

OTHER OUTCOMES:
Compare group difference about stool fermentation production before and after intervention. | Three weeks
  Compare group difference about stool fermentation production- short chain fatty acids, before and after 3-week intervention .
Compare group difference about fecal microbial α- diversity displayed by Shannon index before and after intervention. | Three weeks
  Fresh feces will be collected from patients at baseline and the end of the intervention (three weeks intervention), and the fecal DNA will be extracted by MOBIO PowerSoil DNA Isolation Kit according to the instructions. The 16S rRNA sequencing will be performed from the extracted DNA. Within-community diversity (α- diversity displayed by Shannon index) will be further calculated according to the sequencing results.
Compare group difference about fecal microbial β- diversity displayed by Principal Component Analysis (PCA) before and after intervention. | Three weeks
  Fresh feces will be collected from patients at baseline and the end of the intervention (three weeks intervention), and the fecal DNA will be extracted by MOBIO PowerSoil DNA Isolation Kit according to the instructions. The 16S rRNA sequencing will be performed from the extracted DNA. Between-community diversity (β- diversity displayed by Principal Component Analysis (PCA)) will be further calculated according to the sequencing results.
Compare group difference about fecal microbial communities before and after intervention. | Three weeks
  Fresh feces will be collected from patients at baseline and the end of the intervention (three weeks intervention), and the fecal DNA will be extracted by MOBIO PowerSoil DNA Isolation Kit according to the instructions. The 16S rRNA sequencing will be performed from the extracted DNA. LEfSe (linear discriminant analysis coupled with effect size measurements) will be further calculated according to the sequencing results.
Compare stool microbial α- diversity displayed by Shannon between responders and non-responders | Baseline (0 week)
  Fresh feces collected from responders and nonresponders to interventions at baseline will be analyzed by 16S rRNA sequencing. Within-community diversity (α- diversity displayed by Shannon index) will be further calculated according to the sequencing results.
Compare stool microbial β- diversity displayed by Principal Component Analysis (PCA) between responders and non-responders | Baseline (0 week)
  Fresh feces collected from responders and nonresponders to interventions at baseline will be analyzed by 16S rRNA sequencing. Between-community diversity (β- diversity displayed by Principal Component Analysis (PCA)) will be further calculated according to the sequencing results.
Compare stool microbial communities between responders and non-responders | Baseline (0 week)
  Fresh feces collected from responders and nonresponders to interventions at baseline will be analyzed by 16S rRNA sequencing. LEfSe (linear discriminant analysis coupled with effect size measurements) will be further calculated according to the sequencing results.
Compare stool fermentation production between responders and non-responders | Baseline (0 week)
  Compare stool fermentation production- short chain fatty acids, between responders and non-responders
Compare IBS symptom severity between responders and non-responders | Baseline (0 week)
  Compare IBS symptom severity (measured by IBS symptom severity scale(IBS-SSS)) between responders and non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Yawen Zhang, MM, Principal Investigator — Sir Run Run Shaw Hospital; Lijun Feng, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital , College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang Y, Feng L, Wang X, Fox M, Luo L, Du L, Chen B, Chen X, He H, Zhu S, Hu Z, Chen S, Long Y, Zhu Y, Xu L, Deng Y, Misselwitz B, Lang BM, Yilmaz B, Kim JJ, Owyang C, Dai N. Low fermentable oligosaccharides, disaccharides, monosaccharides, and polyols diet compared with traditional dietary advice for diarrhea-predominant irritable bowel syndrome: a parallel-group, randomized controlled trial with analysis of clinical and microbiological factors associated with patient outcomes. Am J Clin Nutr. 2021 Jun 1;113(6):1531-1545. doi: 10.1093/ajcn/nqab005. PMID 33740048